CLINICAL TRIAL: NCT05374018
Title: Prospective Study to Evaluate Stretococcus Pneumoniae Serotype Prevalence in Community Acquired Pneumonia in Hong Kong Using a Urinary Kit
Brief Title: Urinary Antigen Test for Stretococcus Pneumoniae Serotype Prevalence in Community Acquired Pneumonia
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, To Kin Wang, Prof., Chinese University of Hong Kong
Other Study IDs: CREC 2020.34
Record Dates: First submitted 2022-05-10; First posted 2022-05-13 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: urinary kit for pneumococcus antigen assay — urine test for detection of pneumococcus antigen

SUMMARY:
This is an epidemiology study for the prevalence and serotypes of pneumococcus pneumoniae in hospitalized patients with community acquired pneumonia (CAP). The serotypes of the pneumococcus pneumoniae will be determined by a urinary antigen assay

ELIGIBILITY:
Inclusion Criteria:

Admitted with signs and symptoms suggestive of pneumonia which include one or more of the followings:

1. fever
2. CXR changes with consolidation, increased alveolar shadowing or hazziness
3. respiratory symptoms like increase shortness of breath, cough with sputum Raised inflammatory markers suggesting of bacterial infection with either increased white cell count or C-reactive protein, or both

Exclusion Criteria:

* Nosocomial pneumonia which is acquired >= 48 hours after hospital admission. Pneumonia which are already known to be caused by pathogens other than pneumococcus pneumoniae.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients admitted for CAP
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
prevalence of strep pneumonia | 2 years
  to determine prevalence

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine and Therapeutics, Prince of Wales Hospital, CUHK, Shatin, Hong Kong